CLINICAL TRIAL: NCT07331740
Title: Parenting Concerns of Young and Middle-aged Women With Breast Cancer: A Study Protocol for a Feasibility Trial
Brief Title: Development and Application of a Parenting Anxiety Intervention Program for Young and Middle-Aged Female Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Hu Hanqi, Master's Student, School of Nursing, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: To be assigned
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Parenting Anxiety
Keywords: Young and middle-aged female breast cancer patients; Intervention program; Feasibility trial; Parenting Anxiety
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm feasibility trial; all eligible participants receive the parenting anxiety intervention program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenting Concerns Intervention Group (Experimental): All eligible participants will receive the tailored parenting concerns intervention program.
  Interventions: Behavioral: Parenting Concerns Support Program

INTERVENTIONS:
Behavioral: Parenting Concerns Support Program — A 6-week program including 2 individual psychological counseling sessions and 4 group parenting guidance activities, designed to reduce parenting concerns in young and middle-aged female breast cancer patients.

SUMMARY:
This feasibility study aims to develop and test an intervention program for young and middle-aged female breast cancer patients who experience parenting concerns. Eligible participants will receive the tailored support program (including psychological counseling and parenting guidance). The study will assess whether the program is acceptable, feasible, and potentially helpful in reducing parenting concerns among this group.We plan to enroll 20 participants from Shanghai Zhoupu Hospital between March 2026 and October 2026.

ELIGIBILITY:
Inclusion Criteria:

* Clear breast cancer patients confirmed by histopathology who have received surgical treatment
* Aged 18 to 59 and currently raising at least one minor child under the age of 18
* Clinical stage I - IV
* Be aware of the condition, provide informed consent and voluntarily participate in this study
* The patient can cooperate with the research independently and has normal reading, comprehension, thinking and judgment abilities

Exclusion Criteria:

* Concurrent with other cancers
* Engaged in psychology work, or having received psychological intervention guidance within the past six months
* Participate in other nursing intervention studies simultaneously

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Parenting Concerns Scale for Breast Cancer Patients | Baseline (pre-intervention) , 6 weeks post-intervention (end of the program) and One month after the intervention ended
  This scale was developed by Qian Meiyan et al. in 2024 to assess the parenting anxiety level of breast cancer patients. The scale mainly consists of 5 dimensions and 25 items, namely disease communication (5 items), children's health (4 items), children's emotions (6 items), role communication (6 items), and family support (4 items).

SECONDARY OUTCOMES:
Parenting Sense of Competence Scale | Baseline (pre-intervention), 6 weeks post-intervention (end of the program) and One month after the intervention ended
  This scale was created by Gibaud-Wallston in 1977, aiming to assess the self-perception and confidence level of caregivers.
Herth hope index | Baseline (pre-intervention) , 6 weeks post-intervention (end of the program) and One month after the intervention ended
  Compiled by American scholar Herth in 1991, it is applicable to the survey of hope levels among healthy or sick adults. This scale continues to consist of 3 dimensions and 12 items, namely positive attitudes towards reality and the future, taking positive actions, and maintaining close relationships with others.